CLINICAL TRIAL: NCT02909972
Title: A Phase 1/1b Open-Label Study to Determine the Safety and Tolerability of ALRN-6924 Alone and in Combination With Cytarabine (Ara-C) in Patients With Relapsed/Refractory Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome With Wild-Type TP53
Brief Title: Safety Study of ALRN-6924 in Patients With Acute Myeloid Leukemia or Advanced Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aileron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALRN-6924-1-02
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALRN-6924 (Experimental): Fixed dose of ALRN-6924 per cohort, administered IV, Days 1, 8, and 15 every 28 days
  Interventions: Drug: ALRN-6924
- ALRN-6924 in combination with cytarabine (Experimental): Cytarabine (100 or 200 mg/m2) will be administered as an IV infusion followed by ALRN-6924 on Days 1, 8, and 15 every 28 days.
  Interventions: Drug: ALRN-6924 in combination with cytarabine

INTERVENTIONS:
Drug: ALRN-6924 — Fixed dose of ALRN-6924 per cohort, administered IV, Days 1, 8, and 15 every 28 days.
  Arms: ALRN-6924
Drug: ALRN-6924 in combination with cytarabine — Cytarabine (100 or 200 mg/m2) will be administered as an IV infusion followed by ALRN-6924 on Days 1, 8, and 15 every 28 days.
  Other Names: ALRN-6924 in combination with Ara-C
  Arms: ALRN-6924 in combination with cytarabine

SUMMARY:
Phase 1/1b, open label, multi-center dose escalation and dose expansion study designed to evaluate safety, tolerability, PK (pharmacokinetics), PD (pharmacodynamics) and anti-tumor effects of ALRN-6924 alone or in combination with cytarabine in patients with relapsed/refractory acute myeloid leukemia or advanced myelodysplastic syndrome with wild-type (WT) TP53

DETAILED DESCRIPTION:
Phase I, open label, multi-center dose escalation (DEP) and dose expansion (EXP) study designed to evaluate safety, tolerability, PK (pharmacokinetics), PD (pharmacodynamics) and anti-tumor effects of ALRN-6924 in patients with acute myeloid leukemia or advanced myelodysplastic syndrome with wild-type (WT) TP53. ALRN-6924 is a stabilized cell-permeating peptide designed to disrupt interaction between the p53 tumor suppression protein and its endogenous inhibitors murine double minute 2 (MDM2) and murine double minute X (MDMX)

Men and women 18 years of age and older with relapsed or refractory acute myeloid leukemia or advanced myelodysplastic syndrome and for which standard treatment(s) are not available or are no longer effective can be enrolled. Treatment of patients in the DEP and EXP phases will continue in the study until documentation of disease progression, unacceptable toxicity, or patient or physician decision to discontinue study participation is made.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute myeloid leukemia or IPSS-R intermediate/high/very high-risk MDS patients
* Confirmed or anticipated wild-type TP53
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Adequate hepatic and renal function
* Acceptable coagulation function
* Negative serum or urine pregnancy test within 7 days prior to the first dose of ALRN-6924 for women of child-bearing potential
* Sufficient wash out from prior therapies and recovery from all significant toxicities

Exclusion Criteria:

* Patients are eligible for available approved standard therapies
* Prior treatment with MDM2 inhibitor, with protocol specified exceptions
* Patients with history of allogeneic stem cell transplantation
* Leukemic blast counts of >25,000/µl
* Deletion of chromosome 17, or del(17p)
* Patients with evidence of current central nervous system leukemic involvement
* Known hypersensitivity to any study drug component
* History of coagulopathy
* Prior specified cardiovascular risk factors
* Clinically significant gastrointestinal bleeding within 6 months
* Clinically significant third-space fluid accumulation
* Pregnant or lactating females
* Evidence of any serious and/or unstable pre-existing medical condition that would interfere with patient safety ability to provide informed consent
* Active uncontrolled infection, including HIV/AIDS or Hepatitis B or C
* Second malignancy within one year, with protocol specified exceptions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ALRN-6924 alone and in combination with cytarabine | From Day 1 of treatment until 30 days after the last cycle of treatment (each cycle is 28 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v.4.0
Determine maximum tolerated dose (MTD) | From the first dose until the end of Cycle 2 (each cycle is 28 days)
  Determine the dose limiting toxicities (DLT) and the maximum tolerated dose (MTD) or the optimal biological dose (OBD) of ALRN-6924 in adult patients with AML or MDS

SECONDARY OUTCOMES:
Determine PK parameters of ALRN-6924 when administered to patients with acute myeloid leukemia (AML) or advanced myelodysplastic syndrome (MDS) | First 2 cycles (each cycle is 28 days)
  Peak Plasma Concentration (Cmax)
Determine PK parameters of ALRN-6924 when administered to patients with acute myeloid leukemia (AML) or advanced myelodysplastic syndrome (MDS) | First 2 cycles (each cycle is 28 days)
  Area under the plasma concentration versus time curve [AUC]
Determine immunogenicity of ALRN-6924 | Approximately 16 weeks
  Incidence of anti-ALRN-6924 antibodies
Determine best overall response, duration of response, morphologic leukemia-free state, leukemia free survival, percentage of MDA patients who have achieved hematologic improvement, changes in transfusion rate and early death rate | Approximately 16 weeks
  International Working Group (IWG) Criteria (Cheson et al, 2006)
Determine best overall response, duration of response, morphologic leukemia-free state, leukemia free survival, percentage of MDA patients who have achieved hematologic improvement, changes in transfusion rate and early death rate | Approximately 16 weeks
  AML response criteria (Dohner et al, 2010)
Determine best overall response, duration of response, morphologic leukemia-free state, leukemia free survival, percentage of MDA patients who have achieved hematologic improvement, changes in transfusion rate and early death rate | Approximately 16 weeks
  International Working Group (IWG) Criteria for hematological improvement in MDS (Cheson et al, 2000)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Denver, Colorado
  - Tampa, Florida
  - The Bronx, New York
  - Portland, Oregon
  - Greenville, South Carolina
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No